CLINICAL TRIAL: NCT03079544
Title: Social Media-based Patient Education and Active Self-report on Incidence and Outcomes of Adverse Events in Natural Killer/T-cell Lymphoma (NK/TCL) Patients
Brief Title: Social Media-based Active Self-report on Incidence and Outcomes of Adverse Events in NK/TCL Patients
Status: Completed | Type: Observational
Sponsor: Rong Tao (Other)
Responsible Party: Sponsor-Investigator, Rong Tao, Clinical Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: XHLSG-NK-1603
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Extranodal NK-T-Cell Lymphoma, Nasal Type
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Asparaginase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: L-Asparaginase or or Pegaspargase containing chemotherapy — Patients receive at least one cycle of combinational chemotherapy containing L-asparaginas or Pegaspargase.

SUMMARY:
The purpose of this study is to collect data from patients by social media and self-report on the adverse events and outcomes happened with patients with extranodal natural killer/T-cell lymphoma, nasal type, who are treated outside of clinical trials in China.

DETAILED DESCRIPTION:
Extranodal natural killer/T-cell lymphoma, nasal type, is a rare subtype of non-Hodgkin lymphoma with relatively high incidence in China. L-asparaginase based chemotherapy are widely used with Chinese patients and has been reported to improve overall response and prolonged the long-term survival in some clinical trials with very limited patients. However, most patients were treated out of clinical trials in China. Therefore the real incidence of adverse events and treatment outcomes are largely unknown. This study is designed to evaluate the incidence of adverse events and treatment outcomes by social media-based (www.house086.com, www.wechat.com) self-report from patients who are treated out of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of extranodal natural killer/T-cell lymphoma, nasal type based on WHO 2008 classification of tumors of haematopoietic and lymphoid tissue.
* Treated with at least one cycle of L-asparaginas or Pegaspargase based chemotherapy.
* Signed Informed consent.

Exclusion Criteria:

* patients who are enrolled in any other clinical trials.
* Relapsed patients who were initially treated with non-L-asparaginas or non-pegaspargase based regimens.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with the diagnosis of NK/TCL treated out of clinical trials are candidators for this study.
Sampling Method: Non-Probability Sample
Enrollment: 665 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
overall survival | 2-year
  The overall survial time of patients will be measured since the initiation of treatment to death of any reason.

SECONDARY OUTCOMES:
Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Day 1 of each course of chemotherapy and radiotherapy then every 3 months for 2 years
  Chemotherapy-related and radiotherapy-related toxicities and adverse events will be collected and graded by NCI CTCAE v4.0 criteria.
Progression free survival | 2-year
  Progression free survival time is defined as the time from the initiation of treatment to the date on which disease "progresses" or the date on which the patient dies, from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Study Chair — Xinhua hospital, Shanghai Jiao Tong University of Medicine
Locations (2):
- China (2):
  - Lymphoma House086, Beijing, Beijing Municipality
  - Xinhua Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No